CLINICAL TRIAL: NCT06395909
Title: A Real-World, Retrospective, Multicenter Study to Assess the Effectiveness and Safety of Mayzent® (Siponimod) in Chinese Patients With Relapsing Forms of Multiple Sclerosis
Brief Title: A Study to Assess the Effectiveness and Safety of Mayzent in Chinese Patients With Relapsing Forms of Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: CBAF312A2413
Record Dates: First submitted 2024-04-28; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-05

CONDITIONS: Relapsing Multiple Sclerosis; Clinically Isolated Syndrome; Relapsing Remitting Multiple Sclerosis; Secondary Progressive Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: US Export: Yes

GROUPS / COHORTS (1):
- Siponimod cohort: Patients who were at least 18 years old diagnosed with clinically isolated syndrome (CIS), relapsing-remitting multiple sclerosis (RRMS), or active secondary progressive multiple sclerosis and had received at least 3 months of siponimod treatment after the index date.

SUMMARY:
This was a multicenter, non-interventional, retrospective study aiming to evaluate the real-world effectiveness and safety of siponimod treatment in Chinese patients with relapsing forms of multiple sclerosis (RMS). The data were collected retrospectively through medical records review and abstraction conducted at a single time point per patient by the investigator's site staff or a designate (at the discretion of the site, if allowed by local regulations). There was no prospective patient follow-up for this study. Obtaining informed consent was based on local regulations. Where permissible, waivers could be applied to the Institutional Review Board (IRB) or Independent Ethics Committee (IEC) as appropriate, based on the retrospective collection of non-personally identifiable data, if acceptable per local regulations.

The target patient population included adult patients diagnosed with RMS (including clinically isolated syndrome (CIS), relapsing-remitting multiple sclerosis (RRMS), or active secondary progressive multiple sclerosis (SPMS)), and who received at least 3-months of treatment with siponimod after the index date. The index date is the date of siponimod initiation, defined as the date of first prescription record of siponimod in the patient's medical records with RMS diagnosis. Effectiveness data (i.e., clinical relapses, magnetic resonance imaging (MRI) activity) were collected from the index date, through the end of the observation period. The observation period was from the index date to the date of initiation of medical records abstraction at site, or patient withdrawal of consent, loss of follow-up, or death, whichever occurred first. Among patients who permanently discontinued siponimod during the observation period, safety data were collected up to 30 days after the last dose of siponimod.

ELIGIBILITY:
Inclusion criteria:

* Written informed consent if requested by local regulation.
* Patients had a diagnosis of RMS (including CIS, RRMS, or active SPMS).
* Chinese patients were 18 years or older at the index date.
* Patients had a minimum 3-month persistence on siponimod after the index date.
* Patients had at least one documented clinical visit in the observation period after the initiation of siponimod treatment.

Exclusion criteria:

• Patients previously treated with siponimod (including participation in clinical trials) before the index date.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2023-04-23 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Annualized Relapse Rate (ARR) | Up to approximately 32 months
  The ARR was calculated using the total number of relapses (as documented in the patient's medical records) after index date divided by the total person days of follow-up after index date multiplied by 365.25.

SECONDARY OUTCOMES:
Proportion of Patients Relapse-free at 12 Months after Index Date | 12 months
Proportion of Patients Free of Magnetic Resonance Imaging (MRI) Activity at 12 Months after Index Date | 12 months
Proportion of Patients with Treatment-emergent Adverse Events (TEAEs), per Category | Up to approximately 32 months
  Categories were TEAEs, treatment-related TEAEs, serious TEAEs, TEAEs leading to discontinuation of siponimod, TEAEs leading to death, and TEAEs of special interest (AESIs).
  TEAEs were defined as any AEs that were not presented prior to medical treatment, or an already presented event that worsens either in intensity or frequency following the treatment, that developed after siponimod initiation.
Proportion of Patients with Selected Notable Abnormal Laboratory Data | Up to approximately 32 months
  Selected notable abnormal laboratory data included complete blood count with differential lymphocyte count and liver function tests.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, East Hanover, New Jersey, United States